CLINICAL TRIAL: NCT00740922
Title: A Multicenter Clinical Evaluation of the Safety Follow-up of Becaplermin or Placebo Gel Following Treatment of Chronic, Full Thickness Diabetic Ulcers
Brief Title: Evaluation of the Safety Follow-up of Becaplermin or Placebo Gel Following Treatment of Chronic, Full Thickness Diabetic Ulcers
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Clinical Leader, Internal Medicine, EP, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Other Study IDs: CR004156
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Platelet-Derived Growth Factor; Diabetic Foot; Neoplasms
Keywords: Becaplermin gel; Target Ulcer; Retrospective Studies; Diabetic Foot; Neoplasms; Long-Term Safety; Topical Administration
MeSH Terms: conditions — Diabetic Foot; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Sterile becaplermin gel vs. sterile placebo gel treatment 1

INTERVENTIONS:
Drug: Sterile becaplermin gel vs. sterile placebo gel treatment 1 — Becaplermin gel 100 µg/g versus placebo gel (up to 12 applications).

SUMMARY:
The purpose of this study is to retrospectively evaluate the safety of sterile becaplermin gel compared with sterile placebo gel treatment 12 months or more after the last dose was administered in 1 of 2 double-blind trials [neither the physician nor the patient knows the name of the study drug (PDGF-DBFT-003 and PDGF-DBFT-005].

DETAILED DESCRIPTION:
This single-visit, retrospective study was designed to evaluate the long-term safety of becaplermin gel 100 mcg/g versus placebo gel. Patients previously enrolled in protocol PDGF-DBFT-003 or PDGF-DBFT-005 were evaluated during a single-study visit in which retrospective safety data were collected. Recurrence data on the Target Ulcer were also obtained. The maximum number of patients in this study was the sum of patients enrolled in the 2 previous trials. The investigators made every effort to contact all patients enrolled in the previous double-blind trials in order to get follow-up information on as many patients as possible. If the patient was deceased, the cause of death, if known, was collected by the investigator (where permitted by the local authorities). After evaluation of the entrance criteria, demographic data, significant new intercurrent illnesses, a current medication profile, therapies received for the treatment of any diabetic neuropathic foot ulcer and surgeries in the last 12 or more months were collected and recorded. A questionnaire was used by the investigational staff to elicit patient information. At the visit, a complete physical examination was done (special attention was given to assess the presence of any malignancies), the feet were carefully examined and the footwear was assessed. The site of the Target Ulcer treated in the previous double-blind trial was assessed by an independent dermatologist.and photographs of the heel, back, inside and outside surfaces of the foot, as well as a distance photograph of the foot, were taken. Parameters such as major changes in the general health, (i.e., hospitalizations, major illnesses, and past surgeries), and past as well as present histories of any malignant diseases were carefully assessed. Of primary interest were the examination of previously treated ulcer site(s) and the Target Ulcer limb in general, for recurrences and/or new ulcerations; their treatments and outcomes; and any other relevant changes to the previously treated ulcer and the surrounding skin. Observational study - No study drug administered

ELIGIBILITY:
Inclusion Criteria:

* Patients are required to satisfy the following criteria before entering the study: given written informed consent before the performance of any study-related procedures, if deceased, the cause of death, if known, is collected by the investigator (where permitted by the local authorities)
* Received at least 1 dose of study medication in 1 of the double-blind trials PDGF-DBFT-003 or PDGF-DBFT-005 and had any post-baseline data
* A minimum of 12 months elapsed since last study drug dosing in 1 of the double-blind trials PDGF-DBFT-003 or PDGF-DBFT-005

Exclusion Criteria:

* Patients who meet any of the following criteria are excluded from participating in the study: Patients who are unwilling to participate
* Patients who, despite multiple and documented efforts, could not be contacted (the investigator was asked to try at least 3 times to contact the patient or patient's representative or parents by mail and phone)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic full thickness diabetic ulcers who were treated with becaplermin or placebo gel in two previous studies
Sampling Method: Non-Probability Sample
Enrollment: 563 (Actual)
Dates: Start 1999-07; Study Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to retrospectively evaluate the safety of sterile becaplermin gel vs. sterile placebo gel treatment 12 months or more after the last dose was administered. | single visit 12 months after enrollment

SECONDARY OUTCOMES:
The secondary objective of the trial was to evaluate recurrence of the Target Ulcer if it had healed in the previous trial. | single visit 12 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Evaluation of the safety follow-up of becaplermin or placebo gel following treatment of chronic, full thickness diabetic ulcers. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=558&filename=CR004156_CSR.pdf